CLINICAL TRIAL: NCT00876837
Title: Long-term Outcomes and Life Satisfaction of Adults With Pediatric-Onset Spinal Cord Injuries
Status: Completed | Type: Observational
Sponsor: Shriners Hospitals for Children (Other)
Responsible Party: Principal Investigator, Kathy Zebracki, Director of Psychology, Shriners Hospitals for Children
Other Study IDs: SHC-SCI-LT
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adults with pediatric-onset SCI

SUMMARY:
The purpose of this study is to assess life satisfaction and long-term outcomes (i.e., medical and psychosocial) of adults who sustained spinal cord injuries (SCI) as children or adolescents.

DETAILED DESCRIPTION:
The ultimate goal of rehabilitation for children and adolescents with spinal cord injuries (SCIs) is to assure that they can grow up to have as productive and satisfying lives as their peers. Understanding factors associated with these outcomes of our patients after they have become adults may help to identify interventions and rehabilitation strategies that will optimize long-term outcomes. Long-term studies of adults with pediatric-onset SCI are needed to identify important outcomes, including survival, participation, health status and health-related quality of life, and life-satisfaction. Further, these outcomes need to be compared to population norms. Predictive models of important outcomes will be developed using independent factors, including demographic, impairment, functional limitation, participation, and environmental and personal factors. In addition, the impact of age at injury, upper extremity reconstruction or functional electrical stimulation implants, and the Mitrofanoff procedure on adult outcomes will be assessed. The stability of selected outcomes in comparison to normative and census data will be determined and factors associated with changes in these outcomes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who are 19 years of age and older
* Were injured at the age of 18 years or younger
* Received care at Shriners Hospitals for Children in Chicago, Philadelphia, or Northern California

Exclusion Criteria:

* Non-English speaking individuals due to lack of measures in languages other than English and lack of foreign-speaking research assistants
* severe brain injury

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects for this study are adults who have received care in the SCI Programs of the Shriners Hospitals in Chicago, Philadelphia, or Northern California, who are 19 years of age and older and who were injured at age 18 years or younger.
Sampling Method: Non-Probability Sample
Enrollment: 514 (Actual)
Dates: Start 1998-03; Primary Completion 2020-08-25 (Actual); Study Completion 2020-08-25 (Actual)

PRIMARY OUTCOMES:
medical complications | annually
  Assessment of medical complications, including pressure ulcers, spasticity, UTIs, hospitalizations

SECONDARY OUTCOMES:
psychological outcomes | annually
  assessment of current psychological functioning, including depression, anxiety, happiness, and life satisfaction

OTHER OUTCOMES:
social outcomes | annually
  assessment of social outcomes, including marriage, children, education level, employment status.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Zebracki, Ph.D., Principal Investigator — Shriners Hospitals for Children; Lawrence Vogel, M.D., Principal Investigator — Shriners Hospitals for Children
Locations (1):
- Shriners Hospitals for Children, Chicago, Illinois, United States

REFERENCES:
- [Background] Deane KC, Chlan KM, Vogel LC, Zebracki K. Use of Appraisals of DisAbility Primary and Secondary Scale-Short Form (ADAPSS-sf) in individuals with pediatric-onset spinal cord injury. Spinal Cord. 2020 Mar;58(3):290-297. doi: 10.1038/s41393-019-0375-0. Epub 2019 Nov 7. PMID 31700146
- [Result] Anderson CJ, Vogel LC, Betz RR, Willis KM. Overview of adult outcomes in pediatric-onset spinal cord injuries: implications for transition to adulthood. J Spinal Cord Med. 2004;27 Suppl 1:S98-106. doi: 10.1080/10790268.2004.11753545. PMID 15503711
- [Result] Chen Y, Anderson CJ, Vogel LC, Chlan KM, Betz RR, McDonald CM. Change in life satisfaction of adults with pediatric-onset spinal cord injury. Arch Phys Med Rehabil. 2008 Dec;89(12):2285-92. doi: 10.1016/j.apmr.2008.06.008. PMID 19061740
- [Result] Anderson CJ, Vogel LC, Chlan KM, Betz RR. Coping with spinal cord injury: strategies used by adults who sustained their injuries as children or adolescents. J Spinal Cord Med. 2008;31(3):290-6. doi: 10.1080/10790268.2008.11760725. PMID 18795479
- [Result] Anderson CJ, Vogel LC, Chlan KM, Betz RR, McDonald CM. Depression in adults who sustained spinal cord injuries as children or adolescents. J Spinal Cord Med. 2007;30 Suppl 1(Suppl 1):S76-82. doi: 10.1080/10790268.2007.11754609. PMID 17874691
- [Result] Anderson CJ, Vogel LC, Willis KM, Betz RR. Stability of transition to adulthood among individuals with pediatric-onset spinal cord injuries. J Spinal Cord Med. 2006;29(1):46-56. doi: 10.1080/10790268.2006.11753856. PMID 16572565
- [Result] Vogel LC, Krajci KA, Anderson CJ. Adults with pediatric-onset spinal cord injuries: part 3: impact of medical complications. J Spinal Cord Med. 2002 Winter;25(4):297-305. doi: 10.1080/10790268.2002.11753632. PMID 12482173
- [Result] Anderson CJ, Krajci KA, Vogel LC. Life satisfaction in adults with pediatric-onset spinal cord injuries. J Spinal Cord Med. 2002 Fall;25(3):184-90. doi: 10.1080/10790268.2002.11753620. PMID 12214905
- [Result] Vogel LC, Krajci KA, Anderson CJ. Adults with pediatric-onset spinal cord injury: part 2: musculoskeletal and neurological complications. J Spinal Cord Med. 2002 Summer;25(2):117-23. doi: 10.1080/10790268.2002.11753611. PMID 12137215
- [Result] Vogel LC, Krajci KA, Anderson CJ. Adults with pediatric-onset spinal cord injury: part 1: prevalence of medical complications. J Spinal Cord Med. 2002 Summer;25(2):106-16. doi: 10.1080/10790268.2002.11753610. PMID 12137214
- [Result] Anderson CJ, Vogel LC. Employment outcomes of adults who sustained spinal cord injuries as children or adolescents. Arch Phys Med Rehabil. 2002 Jun;83(6):791-801. doi: 10.1053/apmr.2002.32742. PMID 12048657
- [Result] Zebracki, K., Anderson, C., Chlan, K., & Vogel, L. (2010). Outcomes of adults with pediatric-onset spinal cord injury: Longitudinal findings and implications on transition to adulthood. Topics in Spinal Cord Injury Rehabilitation, 16(1), 17-25. Doi: 10.1310/sci1601-17
- [Result] Vogel LC, Chlan KM, Zebracki K, Anderson CJ. Long-term outcomes of adults with pediatric-onset spinal cord injuries as a function of neurological impairment. J Spinal Cord Med. 2011;34(1):60-6. doi: 10.1179/107902610X12883422813787. PMID 21528628
- [Result] Chlan KM, Zebracki K, Vogel LC. Spirituality and life satisfaction in adults with pediatric-onset spinal cord injury. Spinal Cord. 2011 Mar;49(3):371-5. doi: 10.1038/sc.2010.80. Epub 2010 Jul 6. PMID 20603633
- [Result] Hwang M, Chlan KM, Vogel LC, Zebracki K. Substance use in young adults with pediatric-onset spinal cord injury. Spinal Cord. 2012 Jul;50(7):497-501. doi: 10.1038/sc.2012.8. Epub 2012 Feb 28. PMID 22370762
- [Result] Hwang M, Zebracki K, Chlan KM, Vogel LC. Longitudinal changes in medical complications in adults with pediatric-onset spinal cord injury. J Spinal Cord Med. 2014 Mar;37(2):171-8. doi: 10.1179/2045772313Y.0000000150. Epub 2013 Nov 26. PMID 24090490
- [Result] January AM, Zebracki K, Chlan KM, Vogel LC. Mental health and risk of secondary medical complications in adults with pediatric-onset spinal cord injury. Top Spinal Cord Inj Rehabil. 2014 Winter;20(1):1-12. doi: 10.1310/sci2001-1. PMID 24574817
- [Result] January AM, Zebracki K, Chlan KM, Vogel LC. Symptoms of depression over time in adults with pediatric-onset spinal cord injury. Arch Phys Med Rehabil. 2014 Mar;95(3):447-54. doi: 10.1016/j.apmr.2013.11.011. Epub 2013 Dec 4. PMID 24316327
- [Result] Hwang M, Zebracki K, Chlan KM, Vogel LC. Longitudinal employment outcomes in adults with pediatric-onset spinal cord injury. Spinal Cord. 2014 Jun;52(6):477-82. doi: 10.1038/sc.2014.32. Epub 2014 Mar 25. PMID 24663002
- [Result] Hwang M, Zebracki K, Vogel LC. Occupational characteristics of adults with pediatric-onset spinal cord injury. Top Spinal Cord Inj Rehabil. 2015 Winter;21(1):10-9. doi: 10.1310/sci2101-10. PMID 25762856
- [Result] January AM, Zebracki K, Czworniak A, Chlan KM, Vogel LC. Predictive factors of hospitalization in adults with pediatric-onset SCI: a longitudinal analysis. Spinal Cord. 2015 Apr;53(4):314-9. doi: 10.1038/sc.2015.13. Epub 2015 Feb 10. PMID 25665547
- [Result] Hwang M, Zebracki K, Vogel LC. Medication profile and polypharmacy in adults with pediatric-onset spinal cord injury. Spinal Cord. 2015 Sep;53(9):673-8. doi: 10.1038/sc.2015.62. Epub 2015 Apr 21. PMID 25896344
- [Result] January AM, Zebracki K, Chlan KM, Vogel LC. Sleep, well-being, and psychological symptoms in adults with pediatric-onset spinal cord injury. Rehabil Psychol. 2015 Nov;60(4):328-34. doi: 10.1037/rep0000061. PMID 26618213
- [Result] January AM, Zebracki K, Chlan KM, Vogel LC. Understanding post-traumatic growth following pediatric-onset spinal cord injury: the critical role of coping strategies for facilitating positive psychological outcomes. Dev Med Child Neurol. 2015 Dec;57(12):1143-9. doi: 10.1111/dmcn.12820. Epub 2015 Jun 11. PMID 26095798
- [Result] Murray CB, Zebracki K, Chlan KM, Moss AC, Vogel LC. Medical and psychological factors related to pain in adults with pediatric-onset spinal cord injury: a biopsychosocial model. Spinal Cord. 2017 Apr;55(4):405-410. doi: 10.1038/sc.2016.137. Epub 2016 Sep 27. PMID 27670804
- [Result] Hwang M, Zebracki K, Vogel LC. Long-Term Outcomes and Longitudinal Changes of Neurogenic Bowel Management in Adults With Pediatric-Onset Spinal Cord Injury. Arch Phys Med Rehabil. 2017 Feb;98(2):241-248. doi: 10.1016/j.apmr.2016.07.004. Epub 2016 Jul 26. PMID 27473299
- [Result] January AM, Zebracki K, Chlan KM, Vogel LC. Poor sleep in adults with pediatric-onset spinal cord injury: associations with pain, health, and activity. J Spinal Cord Med. 2017 Sep;40(5):560-566. doi: 10.1080/10790268.2017.1308109. Epub 2017 Apr 10. PMID 28394218
- [Result] January AM, Kirk S, Zebracki K, Chlan KM, Vogel LC. Psychosocial and Health Outcomes of Adults With Violently Acquired Pediatric Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2018 Fall;24(4):363-370. doi: 10.1310/sci17-00012. Epub 2018 Feb 12. PMID 30459499